CLINICAL TRIAL: NCT04241211
Title: Comparative Study for Incidence of Proximal Junctional Kyphosis Between Parathyroid Hormone and Denosumab Following Adult Spinal Deformity Surgery : A Prospective, Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ho-Joong Kim, professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-1901/514-001
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Spine Deformity
MeSH Terms: interventions — Teriparatide; Denosumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Drug: Denosumab Prefilled Syringe [Prolia]
- TP group (Experimental)
  Interventions: Drug: Forsteo

INTERVENTIONS:
Drug: Forsteo — Patients were administered 20mcg of TP (Forsteo) subcutaneously once a day from the day between before 3months to after 3months about surgery.
  Arms: TP group
Drug: Denosumab Prefilled Syringe [Prolia] — Patients were administered 60mg of denosumab (Prolia) subcutaneously once 6months from the day on before 3months to after 3months about surgery.
  Arms: Control group

SUMMARY:
Medical therapy that can lower PJK rates are also being sought. Teriparatide (TP), a recombinant human parathyroid hormone (PTH 1-34), is a bone forming agent mainly used to treat osteoporotic patients with high risk of osteoporotic fracture. There has been reports suggesting protective effect of prophylactic TP to osteoporotic patients receiving ASD surgery concerning PJK.6 Although it had limitations of small sample size and surgical selection bias owing to study design being retrospective. We hypothesized prophylactic TP would act as to reduce the incidence of PJK and therefore reduce PJF and necessity of revision surgeries in patients after ASD correction surgery. Our study can consolidate the beneficial effect of prophylactic TP to patients receiving ASD surgery by reducing the incidence of PJK.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between 50 years to 80 years of age with ASD
2. Multilevel instrumented fusion
3. Cobb angle above 25̊ in coronal plane deformities, Lumbar lordosis below 20̊ in sagittal plane deformities
4. Minimum follow-up of 1 years

Exclusion Criteria:

1. Diagnosis being tumor or infectious condition like Tb spondylitis were excluded
2. Patients with adverse reactions or contraindications to TP were excluded; side effects to TP or bone cancer or metastasis

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PJK | 15months
  PJK prevalance

CONTACTS AND LOCATIONS:
Locations (1):
- Ho joong Kim, Soeul, Sungnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided